CLINICAL TRIAL: NCT00737906
Title: Surgical Reduction of the Inferior Turbinate Using a Coblation® Device for Treatment of Nasal Obstruction: A Prospective, Multi-center Clinical Study
Brief Title: Surgical Reduction of the Inferior Turbinates for Nasal Obstruction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: ArthroCare Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: E-505DHH
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Rhinitis; Inflammation of the Nasal Mucosa; Inflammation of Nasal Tissue
Keywords: Chronic rhinitis; Nasal Obstruction; Nasal Obstruction Symptoms; Failed Medical Management for Nasal Obstruction; Inflammation of the nasal mucosa; Pediatric Turbinate reduction; Coblation; Arthrocare; ENT; Failed Medical Management for Chronic Sinusitis; Turbinate; Inferior Turbinate Hypertrophy; Bilateral Inferior Turbinate Hypertrophy; Turbinate Hypertrophy; Inferior Turbinate; Bilateral Inferior Turbinate
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): Surgical turbinate reduction procedure
  Interventions: Procedure: Surgical turbinate reduction procedure

INTERVENTIONS:
Procedure: Surgical turbinate reduction procedure — Surgical turbinate reduction using the COBLATION device

SUMMARY:
The primary goal of this post-marketing surveillance study is to assess whether surgical turbinate reduction performed using a Coblation® device is associated with reduced nasal obstruction symptoms.

DETAILED DESCRIPTION:
Chronic rhinitis, or inflammation of the nasal mucosa, is one of the most common causes of nasal obstruction in the pediatric population. Chronic rhinitis may result in mucous gland hypertrophy, engorgement of the vascular system and deposition of collagen in the nasal mucosa. These changes occur most prominently in the inferior turbinate, causing enlargement and nasal obstruction. In children, inferior turbinate hypertrophy is associated with a greater degree of nasal obstruction relative to adults because of their small nasal anatomy.

Cases that do not respond to conservative treatments may be considered for one of many surgical procedures, including turbinate excision, submucosal resection, submucosal cautery, laser treatment, cryosurgery, powered microdebridement, or radiofrequency-based ablation. Clinical studies have shown that bipolar radiofrequency-based plasma (Coblation®) devices are capable of creating focal submucosal lesions with minimal or no damage to structures adjacent to the treated area. At present, however, this technique has not been formally evaluated in children. This study will investigate whether surgical turbinate reduction performed using a Coblation device is associated with reduced nasal obstruction symptoms that has failed to improve with other treatment methodologies.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is >=6 and <=17 years old.
2. Patient has had symptoms of nasal obstruction for >=6 months.
3. Patient has nasal obstruction symptoms unresponsive to at least 8 weeks of documented maximum medical management (as described in Section 4.1).
4. Patient has bilateral hypertrophied inferior turbinates without other abnormalities contributing to nasal obstruction (by nasal evaluation and examination).
5. Patient and parent /guardian agree to participate in the clinical study and to complete all required visits and evaluations.
6. Patient (or guardian) must sign IRB approved informed consent form.

Exclusion Criteria:

1. Patient has clinically significant identifiable structural deformities other than turbinate hypertrophy that may contribute to nasal or upper airway obstruction including:

   1. Septal deviation
   2. Concha bullosa
   3. Enlarged adenoids or tonsils (lingual, palatine, or sphenoid)
   4. Nasal polyps
   5. Nasal valve collapse.
2. Patient has been diagnosed with obstructive sleep apnea not originating from the turbinates.
3. Patient has active or chronic upper airway infection that may contribute to nasal obstruction (not including chronic rhinosinusitis).
4. Patient has active coagulation disorder or patient is receiving anti-coagulants, which cannot be safely stopped for 14 days (7 days prior to surgery and 7 days post-surgery).
5. Patient has systemic disease affecting the nasal passage(e.g. Wegener's granulomatosis).
6. Patient is receiving or has received immunotherapy (any type) within 12 months of enrollment.
7. Patient has a nasal septal perforation.
8. Patient has had any previous turbinate surgery.
9. Patient has had any previous nasal surgery.
10. Patient has had any sinus surgery within 6 months of enrollment.
11. Patient has had an adenoidectomy within 3 months of enrollment.
12. Patient is pregnant or potentially pregnant.
13. Patient or caregiver is incapable of understanding or responding to the study questionnaires.
14. Patient is participating in another clinical study during the 12 month enrollment period.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in nasal obstruction symptoms at 6-weeks post surgery as measured using a validated health-related quality of life questionnaire (SN5) compared to nasal obstruction symptoms measured before surgery using the same questionnaire. | 6 weeks, 6 months, 12 months

SECONDARY OUTCOMES:
Morbidity by determining the frequency, type, and severity of any observed adverse events through 12 months following surgical treatment. | Through 12 months
To assess durability of treatment using: a. Self-reported obstructive symptoms measures b. Physical examination measures, d. Blinded evaluation of anterior rhinoscopy images | 6 weeks, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony M Magit, MD, Principal Investigator — Children's Associated Medical Group, San Diego, CA
Locations (5):
- United States (5):
  - Children's Hospital of San Diego, San Diego, California
  - The Children's Hospital, Aurora, Colorado
  - Center for Pediatric ENT, Boynton Beach, Florida
  - Advanced ENT & Allergy, Louisville, Kentucky
  - Pediatric Otolaryngology Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- [Background] Hol MK, Huizing EH. Treatment of inferior turbinate pathology: a review and critical evaluation of the different techniques. Rhinology. 2000 Dec;38(4):157-66. PMID 11190749
- [Background] Chang CW, Ries WR. Surgical treatment of the inferior turbinate: new techniques. Curr Opin Otolaryngol Head Neck Surg. 2004 Feb;12(1):53-7. doi: 10.1097/00020840-200402000-00015. PMID 14712123